CLINICAL TRIAL: NCT05169307
Title: CREST UK: CPX-351 Real-World Effectiveness and Safety Study
Brief Title: CPX-351 Real-World Effectiveness and Safety Study
Status: Completed | Type: Observational
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CREST UK
Record Dates: First submitted 2021-12-13; First posted 2021-12-23 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; CPX-351; Vyxeos liposomal
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — CPX-351

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CPX-351: Adult patients with newly diagnosed, therapy related acute myeloid leukaemia (t-AML) or AML with myelodysplasia-related changes (AML-MRC) who were treated in routine practice with Vyxeos liposomal in the UK.
  Interventions: Drug: CPX-351

INTERVENTIONS:
Drug: CPX-351 — This is a retrospective, non-interventional, observational study. No study drug will be administered in this study.

SUMMARY:
CPX-351 Real World Effectiveness and Safety Study (CREST UK) is a real-world evidence study designed to collect data on the potential benefits and/or risks of Vyxeos liposomal (liposomal daunorubicin/cytarabine; CPX-351) in routine clinical practice in the United Kingdom (UK).

DETAILED DESCRIPTION:
This is a retrospective, non interventional, multi-centre, single arm, observational study designed to assess patients with newly diagnosed, therapy-related acute myeloid leukaemia (t-AML) or acute myeloid leukaemia with myelodysplasia related changes (AML-MRC) who have been treated with Vyxeos liposomal (liposomal daunorubicin/cytarabine; CPX-351) in routine UK clinical practice and managed as per standard local practice.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years at the start of treatment of AML with Vyxeos liposomal
* Pathological diagnosis of t-AML or AML-MRC according to World Health Organization criteria (with at least 20% blasts in the peripheral blood or bone marrow)
* Patient has received at least one infusion of Vyxeos liposomal, prescribed as per the SmPC
* Patient signs an informed consent form or is included in accordance with an informed consent waiver

Exclusion Criteria:

* Treatment with Vyxeos liposomal as part of a clinical trial or managed access program
* Prior treatment intended for induction therapy of AML; only hydroxyurea is permitted for control of blood counts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed, t-AML or AML-MRC who have been treated with Vyxeos liposomal in routine UK clinical practice and managed as per standard local practice will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Number of Participants Achieving Complete Response/Complete Response with Incomplete Platelet or Neutrophil Recovery in Participants With AML Who Were Treated in Routine Practice With Vyxeos Liposomal | First infusion of Vyxeos liposomal (post-August 2018 approval) to inclusion in study, up to approximately 3 years 4 months
Overall Survival in Participants With AML Who Were Treated in Routine Practice With Vyxeos Liposomal | First infusion of Vyxeos liposomal (post-August 2018 approval) to date of death, up to approximately 3 years 4 months

SECONDARY OUTCOMES:
Number of Vyxeos Liposomal Induction and Consolidation Cycles Administered (Inpatient or Outpatient) in Participants With AML Who Were Treated in Routine Practice With Vyxeos Liposomal | First infusion of Vyxeos liposomal (post-August 2018 approval) to inclusion in study, up to approximately 3 years 4 months
Dose Per Cycle of Vyxeos Liposomal Given During Induction and Consolidation Cycles Administered in Participants With AML Who Were Treated in Routine Practice With Vyxeos Liposomal | First infusion of Vyxeos liposomal (post-August 2018 approval) to inclusion in study, up to approximately 3 years 4 months
Percentage of Participants Transferred for Haematopoietic Stem Cell Transplant (HSCT) in Participants With AML Who Were Treated in Routine Practice With Vyxeos Liposomal | First infusion of Vyxeos liposomal (post-August 2018 approval) to inclusion in study, up to approximately 3 years 4 months
Overall Survival in Participants Post-HSCT With AML Who Were Treated in Routine Practice With Vyxeos Liposomal | Date of HSCT to date of death, up to approximately 3 years 4 months
Mean Duration of Hospitalization Stay of Participants With AML Who Were Treated in Routine Practice With Vyxeos Liposomal | First infusion of Vyxeos liposomal (post-August 2018 approval) to inclusion in study, up to approximately 3 years 4 months

CONTACTS AND LOCATIONS:
Locations (15):
- United Kingdom (15):
  - Belfast City Hospital, Belfast
  - Bristol Royal Infirmary, Bristol
  - University Hospitals Derby and Burton, Derby
  - Western General Hospital (Lothian), Edinburgh
  - Royal Devon and Exeter, Exeter
  - The Leeds Teaching Hospitals NHS Trust, Leeds
  - Leicester Royal Infirmary, Leicester
  - University College London Hospitals, London
  - Royal Marsden, London
  - Royal Liverpool/Clatterbridge, Metropolitan Borough of Wirral
  - James Cook University Hospital, Middlesbrough
  - Peterborough Hospital, Peterborough
  - Queen Alexandra Hospital, Portsmouth, Portsmouth
  - Torbay and South Devon, Torquay
  - New Cross Hospital - Wolverhampton, Wolverhampton

IPD SHARING:
Plan to Share IPD: No